CLINICAL TRIAL: NCT02763514
Title: Efficacy Evaluation of 26 Weeks' Dietary Supplementation With DHA- and EPA-enriched Oils on Cognitive Function and Mood in Healthy Adults
Brief Title: The Effects of DHA- and EPA-enriched Oils on Cognitive Function and Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Pronova BioPharma (Industry)
Responsible Party: Principal Investigator, Philippa Jackson, Dr, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 44N3
Record Dates: First submitted 2016-04-20; First posted 2016-05-05 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Cognitive Function

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- DHA-enriched oil (Active Comparator): 3 g PronovaPure 150:500 EE EU
  Interventions: Dietary Supplement: 3 g PronovaPure 150:500 EE EU
- EPA-enriched oil (Active Comparator): 3 g PronovaPure 500:200 EE EU
  Interventions: Dietary Supplement: 3 g PronovaPure 500:200 EE EU
- Placebo (Placebo Comparator): 3 g Olive oil
  Interventions: Dietary Supplement: 3 g Placebo

INTERVENTIONS:
Dietary Supplement: 3 g PronovaPure 150:500 EE EU
  Arms: DHA-enriched oil
Dietary Supplement: 3 g PronovaPure 500:200 EE EU
  Arms: EPA-enriched oil
Dietary Supplement: 3 g Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effects of EPA- and DHA-enriched omega-3 polyunsaturated fatty acid dietary supplements on cognitive function (episodic memory, attention, working memory, executive function), subjective mood, alertness and mental fatigue after 26 weeks daily supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 25 to 49 years inclusive
* Males and females
* Self-report of good health

Exclusion Criteria:

* English is not first language (some of the cognitive tasks have only been validated in native English speakers)
* Habitual consumption of oily fish exceeds one fish meal per week
* Habitual consumption of omega-3 dietary supplements in the previous 6 months
* Habitual use of dietary supplements within the last month (defined as more than 3 consecutive days or 4 days in total; some supplements that do not impact upon cognitive function e.g. garlic, protein, calcium are allowed. Please check with the research team if you are unsure)
* Are a smoker or consume any nicotine replacement products (e.g. chewing gum, e-cigarettes)
* Food allergies or sensitivities to any of the ingredients contained in the investigational product or any other foodstuff
* Pregnant, trying to get pregnant or breast feeding
* Body Mass Index outside of the range 18-35 kg/m2
* High blood pressure (systolic over 159 mm Hg or diastolic over 99 mm Hg)
* Currently taking blood pressure medication
* Currently taking blood thinning medication (e.g. aspirin, warfarin, heparin)
* Have a respiratory disorder that requires regular medication (Note: participants with asthma who only take their medication occasionally/as required are eligible for this study)
* Have frequent migraines that require medication (more than or equal to 1 per month)
* History or current diagnosis of drug/alcohol abuse
* History of kidney or liver disease, or other severe diseases of the gastrointestinal tract (e.g. iron accumulation, iron utilization disorders, hypercalcaemia, hypercalcaemia), that are likely to interfere with metabolism/absorption/secretion of the product under investigation
* History of neurological or psychiatric illness (excluding depressive illness and anxiety)
* History of head trauma
* Sleep disturbances and/or are taking sleep aid medication
* Blood disorders (e.g. anaemia, haemophilia, thrombocytosis)
* Diagnosis of type I or type II diabetes
* Heart disorder, or vascular illness
* Current diagnosis of depression and/or anxiety
* Over- or under-active thyroid
* Chronic gastrointestinal problems (e.g. Inflammatory Bowel Disease, Irritable Bowel Syndrome, celiac disease)
* Any known active infections
* Diagnosed with or may be at risk of having syphilis, hepatitis, the Human T - lymphotropic virus or the Human Immunodeficiency Virus
* Current or past breast cancer diagnosis and/or a mastectomy
* Health condition that would prevent fulfilment of the study requirements
* Currently participating in or in the past 4 weeks participated in other clinical or nutrition intervention studies

Ages: 25 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 337 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Episodic memory | 26 weeks
  An overall score for Episodic memory will be derived by calculating the average score from 6 separate standardised task outcomes (Zimmediate word recall accuracy + Zdelayed word recall accuracy + Zword recognition accuracy + Zpicture recognition accuracy - Zimmediate word recall errors - Zdelayed word recall errors)/6
Subjective fatigue | 26 weeks
  Subjective fatigue will be derived from the Fatigue subscale of the Profile of Mood States questionnaire

SECONDARY OUTCOMES:
Subjective overall mood disturbance | 26 weeks
  Subjective overall mood disturbance is derived from the overall score of the Profile of Mood States questionnaire
Subjective vigour | 26 weeks
  Subjective vigour will be derived from the Vigour subscale of the Profile of Mood States questionnaire
Subjective confusion | 26 weeks
  Subjective confusion will be derived from the Confusion subscale of the Profile of Mood States questionnaire
Subjective anger | 26 weeks
  Subjective anger will be derived from the Anger subscale of the Profile of Mood States questionnaire
Subjective tension | 26 weeks
  Subjective tension will be derived from the Tension subscale of the Profile of Mood States questionnaire
Subjective alertness | 26 weeks
  Subjective alertness will be derived from an Alertness visual analogue scale presented following cognitive task performance
Subjective mental fatigue | 26 weeks
  Subjective mental fatigue will be derived from a Mental Fatigue visual analogue scale presented following cognitive task performance
Numeric Working memory | 26 weeks
  Reaction time (ms)
Numeric Working memory | 26 weeks
  Accuracy (%)
Simple reaction time | 26 weeks
Stroop task | 26 weeks
  Reaction time (ms)
Stroop task | 26 weeks
  Accuracy (%)
Rapid visual information processing | 26 weeks
  Reaction time (ms)
Rapid visual information processing | 26 weeks
  Accuracy (%)
Verbal fluency | 26 weeks
  Number correct

OTHER OUTCOMES:
Omega-3 index | 26 weeks
  Omega-3 index is expressed as the sum of EPA and DHA as a percentage of total red blood cell fatty acids

CONTACTS AND LOCATIONS:
Overall Officials: Philippa Jackson, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patan MJ, Kennedy DO, Husberg C, Hustvedt SO, Calder PC, Khan J, Forster J, Jackson PA. Supplementation with oil rich in eicosapentaenoic acid, but not in docosahexaenoic acid, improves global cognitive function in healthy, young adults: results from randomized controlled trials. Am J Clin Nutr. 2021 Sep 1;114(3):914-924. doi: 10.1093/ajcn/nqab174. PMID 34113957